CLINICAL TRIAL: NCT00170404
Title: Nutrition, Immunology, and Epidemiology of Tuberculosis
Brief Title: TB Nutrition, Immunology and Epidemiology
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-032
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-02

CONDITIONS: Mycobacterium Tuberculosis
Keywords: HIV Infections, Tuberculosis, Malnutrition, Tanzania
MeSH Terms: conditions — HIV Infections; Tuberculosis; Malnutrition | interventions — Folic Acid; Niacin; Vitamin B 12; Selenium; Vitamin A

INTERVENTIONS:
Drug: Folic Acid
Drug: Micronutrients: Vitamins B1, B2, B6, Niacin, B12, C, E.
Drug: Selenium
Drug: Vitamin A

SUMMARY:
The purpose of this study is to see whether people who take vitamins along with the standard medicine for tuberculosis (TB) recover better and quicker than people who take only the standard medicine for TB. This study will enroll 600 men and women, who are age 18-65 years, have TB, and intend to stay in Dar-es-Salaam for at least 2 years from the start of TB therapy. Half the participants will have active TB and also HIV infection, and the other half will have TB alone. Half the volunteers will be given vitamins, and the other half will be given placebo (sugar pill with no vitamins) from the start of their TB therapy, through the 8 months of anti-TB therapy, and up to 48 months. Participation in the study involves visits to the clinic, physical exams, home visits, and answering questions about personal health, foods eaten, household, occupation, and education. Volunteers will also provide blood, sputum, and urine samples.

DETAILED DESCRIPTION:
This double blinded, randomized, placebo controlled trial will enroll 600 men and women, who are age 18 to 65 years inclusive, have at least two positive sputum smears for tuberculosis (TB), intend to stay in Dar-es-Salaam (DSM) for at least 2 years from the start of TB therapy, and have given informed consent to participate in the study. Half of the enrollees will have active TB and co-infection with HIV, and the other half will have TB alone. The effect of micronutrient status will be examined in the context of a randomized trial conducted in Tanzania. Subjects will be randomized to receive either multi-micronutrients or placebo from the start of their TB therapy, through the 8 months of anti-TB therapy, and until the last recruited patient reaches 24 months of follow up. Thus, the first subject is likely to be followed for 48 months, assuming the duration of recruitment is 24 months. The endpoints of interest include bacteriologic cure, immune response parameters, and clinical outcomes. The researchers will also examine the utility of these immune response parameters as surrogate markers for treatment efficacy in TB, irrespective of nutritional and other risk factors. The study will be carried out as a collaborative effort between Harvard School of Public Health; Muhimbili University College of Health Sciences, Dar es Salaam, Tanzania; Tufts University, Boston; and the Channing Laboratory, Boston. Subjects will be randomly assigned to receive a daily oral dose of one of two treatments: (a) micronutrients: 5000 IU of retinol, 20 mg of B1, 20 mg of B2, 25 mg of B6, 100 mg of niacin, 50 mcg of B12, 500 of C, 200 mg of E, 0.8 mg of folic acid, and 100 mcg of selenium; or (b) placebo. The primary objectives are to: (1) determine the efficacy of micronutrient supplements on sputum and culture negativity at one month and two months; (2) determine the efficacy of micronutrient supplements on survival between two arms at 8 and 24 months; and (3) determine the efficacy of micronutrient supplements on TB relapse and reinfection. Secondary study objectives are to: (1) compare the treatment arms with respect to rate of change of HIV viral load in HIV positive subjects measured at 0, 2, 8, and 20 months; (2) compare the treatment arms with respect to absolute change in CD4 counts from 0 to 2, 8, 20 months; (3) compare the treatment arms with respect to weight change from baseline and 2 months, 8 months, and 20 months; (4) compare the treatment arms with respect to immunological parameters, namely ex vivo lymphocyte proliferation; and cytokine production, namely IL-2, INF-g, IL-12, and TNF-a, at 2, 8, 20 months; and (5) correlate the above mentioned immunological markers with smear conversion rates at 1 month, 2 months, cure, relapse, and death.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 18 to 65 years inclusive
2. At least two positive sputum smears for tuberculosis (TB)
3. Intention to stay in Dar-es-Salaam for at least 2 years after the start of TB therapy
4. Subjects who grant informed consent to participation
5. Subject is assigned to a treatment clinic where International Collarborations in Infectious Disease Research (ICIDR) staff can follow that patient, either at that clinic directly, or through referral to a nearby clinic for research visits.

Exclusion Criteria:

1. Karnofsky score < 40%
2. Hemoglobin < 8.5 g/dl
3. Having had treatment for TB exceeding 4 weeks in the last 5 years
4. Pregnant women: Women who are pregnant at the time of enrollment will also be excluded, given that all pregnant women receive folate and iron supplements as part of routine prenatal services. Also, it is not possible to enroll enough pregnant women to examine the effect of the supplements in this subset.
5. Patient is mentally incapable of understanding the consent form; patient is a prisoner or in police custody; or patient is deaf/dumb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 887
Dates: Start 2000-06; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University, College of Health Sciences, Dar es Salaam, Tanzania